CLINICAL TRIAL: NCT02934880
Title: Study of Impact of Adapted Physical Activity on Cognitive Functions and Quality of Life in Patients Treated for Locally Advanced Breast Cancer
Brief Title: Impact of Adapted Physical Activity on Cognitive Functions in Breast Cancer
Acronym: COG-SPORTIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHB16.01
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: adapted physical activity, cognitive functions
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate APA (Experimental): intervention: 10 sessions of APA within the 5 weeks (2 sessions per week) following the randomization
  Interventions: Other: immediate APA program
- Delayed APA (Active Comparator): intervention: 10 sessions of APA in 5 weeks (2 sessions per week) , 3 months after randomization
  Interventions: Other: delayed APA program

INTERVENTIONS:
Other: immediate APA program — 10 sessions of one hour APA in 5 weeks after patient randomization. 2 sessions per week will be organized
  Arms: Immediate APA
Other: delayed APA program — 10 sessions of one hour APA in 5 weeks 3 months after patient randomization. 2 sessions per week will be organized
  Arms: Delayed APA

SUMMARY:
Breast cancer is the most frequent cancer in women in western countries. The improvement of therapeutic management associated to the developement of supportive care allows patient to live longer in better conditions. But several studies have showed the deleterious impact of treatment such as chemotherapy on cognition. To limit these damages, non therapeutic approaches such as Adapted Physical Activity (APA) have been developped.

The goal of this study is to evaluate the benefit of APA program on cognitive functions in patients with locally advanced breast cancer.

DETAILED DESCRIPTION:
Patient with cognitive complaint will be randomized in two groups :

* Experimental group : Immediate APA program (after randomization)
* Standard group : Delayed APA program (3 months after randomization)

APA program contains 10 sessions of APA within five weeks (twice a week). Each session is composed of 5 exercises (each made of 3 serial of 7 repetitions in slow speed).

A cognitive and quality of life assessments will occur in two groups at 3 and 6 months after randomization.

The primary objective of the study is to evaluate the impact of APA program on the improvement of cognitive functions in patients with breast cancer who have been treated by adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Women
* More than 18 years old
* Locally advanced breast cancer
* Patient who undergone surgery
* Cognitive complaint (FACT-COG inferior or equal to 8/16)
* No metastasis at the inclusion
* Patient who received adjuvant therapy by chemotherapy
* Patient with a social protection
* Barbizet scale Superior or equal to 3
* No neurological history
* No medical contraindication to APA
* Inform consent signed

Exclusion Criteria:

* Metastatic breast cancer
* History of other cancer (in 5 years before inclusion)
* Current chemotherapy or radiotherapy
* Chemotherapy or radiotherapy ended for more than 6 months
* Current APA program
* Blood transfusion for less than 6 mois
* Minimal mental score inferior to normal
* Patient no able to respond to the cognitive test
* Patient no able to realize APA program
* Drug use
* Alcohol abuse
* Patient Under guardianship or curatorship or deprived of liberty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
proportion of patient with an increase of Functional Assessment of Cancer Therapy-Cognitive Function (FACT-COG) result | After APA program
  Proportion of patient with an increase superior or equal to seven points between FACT-COG at the inclusion and FACT-COG after APA program

SECONDARY OUTCOMES:
Improval of quality of life | After APA program
  Impact of APA on quality of life (FACT-B result)
Comparison of immediate APA and delayed APA on quality of life | 30 months
  Comparison between FACT-B, FACT-COG and FACIT-F results in the two groups
Study of relations between cognitive functions and quality pf life | After APA program
  Correlation between patient questionnaire and data of psychological tests done by neuropsychologist

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rigal, MD, Principal Investigator — Centre Henri Becquerel
Locations (3):
- France (3):
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No